CLINICAL TRIAL: NCT00420121
Title: European Society of Cutaneous Lupus Erythematosus
Brief Title: European Society of Cutaneous Lupus Erythematosus (EUSCLE)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: European Society of Cutaneous Lupus Erythematosus e.V. (Other)
Responsible Party: Principal Investigator, Prof. Dr. Annegret Kuhn, Professor, European Society of Cutaneous Lupus Erythematosus e.V.
Other Study IDs: 2742-2
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic
Keywords: standardized evaluation; core set questionnaire; epidemiological data; laboratory analysis
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: laboratory analysis — blood withdrawal for laboratory analysis

SUMMARY:
Cutaneous lupus erythematosus (CLE) is a disease with a wide spectrum of clinical manifestations and a variable prognosis. The aim of the study is to create a standardized evaluation of the different subtypes of this disease in order to receive an overview of the spectrum of clinical and laboratory features as well as the therapeutic strategies for patients with CLE.

DETAILED DESCRIPTION:
Methods: A core set questionnaire has been developed in the course of the "European Society of Cutaneous Lupus Erythematosus (EUSCLE)", and a total of 40 patients (32 females, 8 males) in two centres, Germany and Sweden, were included in this study. Results: CLE was diagnosed in 39 individuals (5 with acute CLE, 10 with subacute CLE, 13 with chronic CLE, and 18 with intermittent CLE) and one individual presented with a systemic manifestation of the disease. Furthermore, disease onset and duration as well as activity and damage of skin lesions using a modified CLASI were examined. Interestingly, 75% of the patients with CLE showed a positive history of photosensitivity, but only 62.5% exhibited characteristic lesions after standardized phototesting. Laboratory analysis revealed positive antinuclear antibodies in 50% of the patients, positive anti-Ro/SSA in 12 and positive anti-La/SSB antibodies in 8 cases. The predominantly used treatments included sunscreens (38 patients), topical steroids (31 patients), topical calcineurin inhibitors (12 patients), chloroquine (19 patients), hydroxychloroquine (11 patients), and systemic steroids (12 patients). Conclusions: The new core set questionnaire enables the clinician to characterize the different skin manifestations involved in CLE and to evaluate disease activity and reasonable treatment modalities. Furthermore, epidemiological data and laboratory features can be assessed for the various subtypes. In the future, this standardized evaluation might lead to the development of diagnostic guidelines and evidence based therapeutic strategies thus improving quality of care for patients with CLE.

ELIGIBILITY:
Inclusion Criteria:

* systemic or cutaneous lupus erythematosus confirmed by histological analysis
* written informed consent available prior to any study-procedures

Exclusion Criteria:

* patients with conditions that are contrary to the above mentioned criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic or cutaneous lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-01; Primary Completion 2018-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Activity and Damage of Skin Lesions in Patients with Cutaneous Lupus Erythematosus measured by the RCLASI Activity and Damage Score. | Up to 12 months
  The Total RCLASI Activity Score measures (i) the activity of skin lesions by evaluating the parameters "erythema", "scaling ⁄hyperkeratosis", "oedema ⁄Infiltration", and "subcutaneous nodule ⁄plaque" and/or (ii) the activity of mucous membrane lesions and/or (iii) the activity of alopecia.
  The Total RCLASI Damage Score measures (i) the damage of skin lesions by evaluating the parameters "dyspigmentation" and "scarring/atrophy" and/or (ii) the damage of scarring alopecia.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, MD, Principal Investigator — University of Muenster, Department of Dermatology
Locations (1):
- University of Muenster, Department of Dermatology, Münster, North Rhine-Westphalia, Germany